CLINICAL TRIAL: NCT03054207
Title: Impact of Antiretroviral Treatment on Pharmacokinetics and Pharmacodynamics of Thienopyridines in Healthy Volunteers and HIV Patients
Acronym: IMPACT/R
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: difficulty to recruit
Sponsor: Jules Desmeules (Other)
Responsible Party: Sponsor-Investigator, Jules Desmeules, Professor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-096
Record Dates: First submitted 2017-02-06; First posted 2017-02-15 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-02

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Clopidogrel; Tablets; Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- HIV clopidogrel (Experimental): clopidogrel 300 mg single dose oral route
  Interventions: Drug: Clopidogrel 300Mg Tablet
- HIV prasugrel (Experimental): prasugrel 60 mg single dose oral route
  Interventions: Drug: Prasugrel 60Mg
- Control clopidogrel (Active Comparator): clopidogrel 300 mg single dose oral route
  Interventions: Drug: Clopidogrel 300Mg Tablet
- Control prasugrel (Active Comparator): prasugrel 60 mg single dose oral route
  Interventions: Drug: Prasugrel 60Mg

INTERVENTIONS:
Drug: Clopidogrel 300Mg Tablet
  Arms: Control clopidogrel; HIV clopidogrel
Drug: Prasugrel 60Mg
  Arms: Control prasugrel; HIV prasugrel

SUMMARY:
HIV patients are at particular risk to develop cardiovascular disease (CVD) as they exhibit multiple risk factors by the nature of their pathology. In addition, the long term exposition to antiretroviral drugs has been associated to an increased risk for CVD. HIV patients can thus potentially receive antiplatelet therapy concomitantly with their antiretroviral treatment. Clopidogrel and prasugrel are thienopyridine antiplatelet agents indicated to prevent the recurrence of ischemic events after coronary arteries stenting. These pro-drugs are mainly bioactivated by cytochromes P450 (CYP) 3A and 2B6 for prasugrel and CYP2C19, CYP3A and CYP2B6 for clopidogrel. Ritonavir is commonly used to "boost" the bioavailability of other HIV drugs through inhibition of CYP3A4 as well as CYP2B6 and CYP2C9. This interaction could therefore reduce clopidogrel and prasugrel efficacy by reducing the formation of their active metabolites. The aim of the present study is to assess the potential drug-drug interaction between clopidogrel/prasugrel and ritonavir. Two groups of 12 male subjects will be constituted (12 HIV patients under ritonavir boosted therapy and 12 healthy volunteers) in a randomized cross-over clinical trial. All subjects will also be genotyped for the CYP2C19. The pharmacokinetics of clopidogrel active metabolite and prasugrel active metabolite will be assessed. Furthermore, the pharmacodynamic response will be evaluated by two gold standard platelet inhibition tests, namely VAsodilator-Stimulated Phosphoprotein Assay (VASP) and VerifyNow® assays. The primary endpoint of this study is to compare the pharmacodynamic response to clopidogrel and prasugrel in HIV patients to that of healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males >18 years
* Understanding of French language and able to give an inform consent
* Anti-HIV therapy with ritonavir or cobicistat (for HIV group)
* Stable antiretroviral treatment since at least 2 weeks (for HIV group)
* Viremia <100 copies/ml (for HIV group)

Exclusion Criteria:

* renal failure: calculated creatinine Clearance (cockcroft) < 50ml/min
* hepatic impairment (ASAT, ALAT, bilirubin, gamma-GT more than 2-fold increase)
* smoker >1 pack/day
* hypersensitivity to any of the drugs used
* intake of any drug or particular food (grapefruit) that can affect CYP activities inhibitors (in the last 10 days before the start of the study or 4 half-life after the last intake)
* pathologies or drugs associated with an increased bleeding risk such as aspirin, non-steroidal anti-inflammatory drugs, steroids and serotonin reuptake inhibitors (in the last 10 days before the start of the study or 4 half-life after the last intake)
* bleeding familial history or antecedent or haemorrhagic disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-06; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Comparison of Platelet Reactivity Index between HIV patients and healthy volunteers | 4hr
  assess the effect of antiretroviral therapies on the response to antiplatelet treatment

SECONDARY OUTCOMES:
Comparison of platelet inhibition between HIV patients and healthy volunteers | 4hr
Comparison of AUC of plasmatic concentrations of prasugrel and clopidogrel between HIV patients and healthy volunteers | 4 hr
Comparison of Cmax of prasugrel and clopidogrel between HIV patients and healthy volunteers | 4 hr
Comparison of Tmax of plasmatic concentrations of prasugrel and clopidogrelpatients and healthy between HIV patients and healthy volunteersvolunteers | 4 hr
Comparison of Half life of prasugrel and clopidogrel between HIV patients and healthy volunteers | 4 hr
Comparison of Clearance of prasugrel and clopidogrel between HIV patients and healthy volunteers | 4 hr

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No